CLINICAL TRIAL: NCT06048432
Title: Effect of Tele-physiotherapy on Patients With Post-stroke Hemiplegia During covid19 Lockdown
Brief Title: Tele-physiotherapy on Post-stroke Hemiplegia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Collaborators: Hermanas Hospitalarias del Sagrado Corazón de Jesús (Unknown); Hospital Universitario Virgen de la Arrixaca (Other)
Responsible Party: Principal Investigator, Juan Jose Hernández Morante, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TELEFISIO-ON-COVID
Record Dates: First submitted 2022-08-07; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Hemiplegia; Muscle Spasticity
Keywords: hemiplegia; stroke; telephyisiotherapy; older adults
MeSH Terms: conditions — Hemiplegia; Muscle Spasticity; Stroke

STUDY DESIGN:
Intervention Model Description: Two groups of patients with post-stroke hemiplegia will be treated only with conventional physiotherapy (CONTROL) or with physiotherapy plus telecare (INTERVENTION).
Who Masked: Participant, Care Provider
Masking Description: Two groups of patients with post-stroke hemiplegia will be treated only with conventional physiotherapy or with physiotherapy plus telecare.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Conventional phyisiotherapy + telecare
  Interventions: Other: Conventional Physiotherapy + telephysiotherapty
- Control (Active Comparator): Conventional physiotherapy
  Interventions: Other: Conventional Physiotherapy + telephysiotherapty

INTERVENTIONS:
Other: Conventional Physiotherapy + telephysiotherapty — Patients assigned to the telephyisiotherapy (TP) group will carry out a half-hour session of conventional therapy, plus a 1-hour session of physical exercise, which will be carried out through the administration of tutorial videos, telephone instructions or by email.

SUMMARY:
The present preliminary randomized trial will be performed to compare the effectiveness of telephyisiotherapy plus physical exercises versus other conventional techniques (electromyographic biofeedback or conventional physiotherapy).

Participants will be chosen from Hospital Sagrado Corazón de Málaga, after the approval of the centre. One hundred and twenty patients with hemiplegia as a consequence of an ischaemic stroke will take part in the study. Selection criteria included to be older than 65 years, with two months of evolution after the stroke and with the left paretic side. In addition, they had to have a positive diagnosis of COVID-19. Positive cases will be confirmed by PCR. Due to the local sanitary regulations, all patients may require home confinement during 1 month without possibility to continue their rehabilitation program.

Physiological interventions started 20 days after the first negative PCR test.

Participants will be randomize in three different intervention groups, conventional therapy (n=40), carried out in the Hospital, biofeedback therapy (n=40), also conducted in the Hospital, and Telephyisiotherapy (TP) plus physical activity (n=40). The intervention period will last for three months, and participants will be re-evaluated 30 days later to confirm treatment effectiveness.

Measurements

Electromyographic activity and hand strength The mean electromyographic (EMG) activity will be determined with the Neurotrans Myoplus 2 Pro System (Verity Medical Ltd, UK), the same instrument used to carry out the intervention. The isometric strength (Nw) of the hand will be assessed with a hand-held digital dynamometer (Smedley digital hand dynamometer, RMS Ltd., UK).

Functional tests In the present work, the Fugl-Meyer will be used to determine the functional status of patients with stroke. The patients with better functionality had superior scores. In addition, the ability of the patients to perform basic daily living activities was determined through the Barthel index. Considering the advanced age of the participants, three extra-scales will be determined: the FRAIL scale, the short physical performance battery (SPPB) and the Strength, assistance in walking, rise from a chair, climb stairs and falls (SARC-F) scale will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hemiplegia as a consequence of an ischaemic stroke
* To be older than 65 years
* Voluntarily participate in the study

Exclusion Criteria:

* To suffer from dementia or severe cognitive decline
* To have any specific contraindication for sport practice (as suffering from joint pain, etc.)
* Those with any diagnosis of severe pathology (cancer, cardiovascular event, etc.) during the study period.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Changes in muscle activity | Determinations will be done through study completion, an average of 1 year.
  Main outcome will be changes in electromyogrpahic activity. A change of plus 10 microvolts will be considered as an effective intervention.

SECONDARY OUTCOMES:
Fugl-Meyer test score | Determinations will be done through study completion, an average of 1 year
  Changes in the specific functional capacity of stroke patients will be determined by the Fugl-Meyer test. A change greater than 10% will be considered beneficial. The Fugl-Meyer test score ranges from 0-66. Higher scores represent better functionality (further information at: PMID: 1135616).

CONTACTS AND LOCATIONS:
Overall Officials: Juan José Hernández Morante, PhD, Principal Investigator — Universidad Católica San Antonio de Murcia
Locations (1):
- Catholic University of Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD will be posted online in a public repository
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Gamez AB, Hernandez Morante JJ, Martinez Gil JL, Esparza F, Martinez CM. The effect of surface electromyography biofeedback on the activity of extensor and dorsiflexor muscles in elderly adults: a randomized trial. Sci Rep. 2019 Sep 11;9(1):13153. doi: 10.1038/s41598-019-49720-x. PMID 31511629
- [Background] Gamez Santiago AB, Martinez Caceres CM, Hernandez-Morante JJ. Effectiveness of Intensively Applied Mirror Therapy in Older Patients with Post-Stroke Hemiplegia: A Preliminary Trial. Eur Neurol. 2022;85(4):291-299. doi: 10.1159/000522413. Epub 2022 Apr 4. PMID 35378544